CLINICAL TRIAL: NCT00869466
Title: B- AHEAD Study (Breast - Activity & Healthy Eating After Diagnosis) Randomised Comparison of 3 Weight Control Programmes During Adjuvant Treatment for Early Breast Cancer.
Brief Title: Weight Control Programs in Women Who Have Undergone Surgery for Early Stage Breast Cancer
Status: Completed | Type: Observational
Sponsor: Wythenshawe Hospital (Other)
Organization: National Cancer Institute (NCI) (NIH)
Other Study IDs: NCGPC-B-AHEAD; CDR0000633348 (Registry Identifier: PDQ (Physician Data Query)); EU-20906
Record Dates: First submitted 2009-03-25; First posted 2009-03-26 (Estimated); Last update posted 2013-04-04 (Estimated); Status verified 2009-03

CONDITIONS: Breast Cancer; Weight Changes
Keywords: weight changes; stage IA breast cancer; stage IB breast cancer; stage II breast cancer; stage IIIA breast cancer; stage IIIB breast cancer; stage IIIC breast cancer
MeSH Terms: conditions — Breast Neoplasms; Body Weight Changes | interventions — Counseling; Early Intervention, Educational

INTERVENTIONS:
Behavioral: behavioral dietary intervention
Behavioral: exercise intervention
Other: counseling intervention
Other: educational intervention
Other: laboratory biomarker analysis
Other: questionnaire administration
Procedure: quality-of-life assessment
Procedure: support group therapy

SUMMARY:
RATIONALE: Measuring changes in body weight and body composition in women with early-stage breast cancer may help doctors plan the best weight control program and improve patients' quality of life. It is not yet known which program is most effective in women with breast cancer.

PURPOSE: This randomized clinical trial is comparing three weight control programs to see how well they work in women who have undergone surgery for early stage breast cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* To assess changes in body weight and composition (i.e., body fat, fat-free mass, dual energy x-ray absorptiometry, bioelectrical impedance, and waist and hip circumference) in patients with early stage breast cancer.

Secondary

* To assess uptake and retention to the interventions and adverse effects of the interventions in these patients.

OUTLINE: This is a multicenter study.

Patients are stratified according to adjuvant treatment (chemotherapy vs no chemotherapy), body mass index (> 27kg/m² vs < 27 kg/m²), treating hospital (UHSM vs North Manchester vs Royal Oldham vs Stepping Hill Hospital), high vs low risk of reducing bone density (i.e., patients receiving aromatase inhibitors vs premenopausal women receiving chemotherapy and/or tamoxifen vs postmenopausal women receiving tamoxifen), and high vs low risk of developing lymphedema (i.e., axillary node clearance vs no axillary node clearance). Patients are randomized to 1 of 3 interventions.

* Arm I: Patients receive standard written advice "Healthy Living With Breast Cancer" booklet from South Manchester University Hospital.
* Arm II: Patients receive individualized diet and exercise advice from a study dietitian for 40 minutes and from the exercise referral officer for 40 minutes. Advice is reinforced with 20-minute bi-weekly phone calls checking compliance, changes in diet, physical activity, individual problems and goals, and recommendations. Patients also receive mailed information summarizing key motivational, behavioral, diet, and exercise issues; information covered in group sessions on weight management; and a booklet providing a program of walking, strengthening, toning, and flexibility exercises.
* Arm III: Patients undergo a supervised group community weight control intervention based on Courneya's exercise prescription guidelines for breast cancer patients and survivors. The intervention consists of a 5-minute warm-up comprising walking and movement to music, 20-30 minutes of circuit training with approximately 10 stations incorporating aerobic activities (i.e., brisk walking, cycling, low-level exercise to music) and muscle strengthening activities (i.e., wall press-up, side leg raises, light weights, and resistance bands), 10-minute cool-down with stretch and flexibility exercises, and 5-minute relaxation period. Patients also undergo a 30-minute diet and behavior change educational session based on the trans theoretical model of behavior changes. The intervention repeats once weekly for 12 weeks. Patients receive a booklet providing a program of walking, strengthening, toning, and flexibility exercises. Patients also receive booster phone calls to reinforce advice, problem solve, and monitor compliance at 4, 6, and 9 months.

In all arms, quality of life is assessed at baseline and 3, 6, and 12 months. Serum bone markers, insulin, glucose, and cardiovascular disease markers are measured periodically.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Diagnosis of early breast cancer

  * Stage I-III disease
  * Invasive or in situ disease
* No metastatic or inoperable disease
* Underwent primary surgery for primary breast cancer at UHSM, North Manchester, Royal Oldham, Stepping Hill, Hope Macclesfield General, Tameside General, Leighton Hospitals, or Rochdale Infirmary within the past 10 weeks
* Receiving/due to start adjuvant chemotherapy, radiotherapy, endocrine therapy, or no adjuvant treatment
* Hormonal receptor status not specified

PATIENT CHARACTERISTICS:

* Pre or postmenopausal status
* Any weight allowed
* Resident within Greater Manchester or Cheshire area
* No physical/psychiatric condition that impairs compliance or mobility as assessed from medical history or baseline fitness assessment, including any of the following:

  * Insulin-requiring diabetes (non-insulin requiring diabetics are eligible)
  * Serious digestive and/or absorptive problems, including inflammatory bowel disease
  * Cardiovascular or respiratory disease
  * Musculoskeletal disease or joint problems
  * Psychiatric disorders or conditions (e.g., untreated major depression, psychosis, substance abuse, or severe personality disorder)
* Not considering reconstructive surgery in the next 12 months

PRIOR CONCURRENT THERAPY:

* See Disease Characteristics
* No concurrent daily medication known to affect body composition (e.g., corticosteroids)

  * Patients receiving 2-3 days of steroids with chemotherapy are eligible
* No prior neoadjuvant chemotherapy or endocrine therapy

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 409 (Actual)
Dates: Start 2008-08; Study Completion 2011-02 (Actual)

PRIMARY OUTCOMES:
Changes in body weight and composition (i.e., body fat, fat-free mass, dual energy x-ray absorptiometry, bioelectrical impedance, and waist and hip circumference) at baseline and at 6 and 12 months

SECONDARY OUTCOMES:
Uptake and retention of information about the interventions and adverse effects of the interventions
Changes in quality of life as assessed by FACT-B, B-ES, and -F at baseline and at 6 and 12 months
Changes in markers of breast cancer prognosis at baseline and at 6 and 12 months
Changes in insulin resistance and glucose homeostasis model assessment (HOMA) at baseline and at 6 and 12 months
Cardiovascular disease-risk markers (i.e., total LDL and HDL cholesterol, triglycerides, and systolic/diastolic blood pressure) at baseline and at 6 and 12 months
Changes in fitness as assessed by a 12-minute walk test at baseline and at 6 and 12 months
Changes in arm mobility, function (as assessed by quick DASH), and pain (as assessed by pain rating scale and S-LANSS for neuropathic pain) at baseline and at 6 and 12 months
Changes in dietary intake (as assessed by a 7-day food diary) and activity (as assessed by a 7-day activity diary) as measures of compliance at baseline and at 6 and 12 months
Changes in serum bone markers/bone specific alkaline phosphatase for bone formation and the cross linked C-telopeptides of type I collagen for bone resorption at baseline and at 6 and 12 months
Changes in ipsilateral arm circumference (compared to contralateral arm) using perometer in patients having axillary node clearance at baseline and at 6 and 12 months
Changes in generic health status and quality of life (as assessed by EQ-5D utility measure) and health resource usage to assess the relative cost effectiveness of the interventions at baseline and at 3, 6, and 12 months
Changes in isometric and isokinetic muscle strength of quadriceps in patients receiving aromatase inhibitors and age-matched patients receiving tamoxifen in a subset of patients in the standard written only group
Patient experience of interventions through in-depth focus group discussions and individual interviews
Factors predicting adherence to interventions with scales of stage of behavior change for weight control and exercise

CONTACTS AND LOCATIONS:
Overall Officials: Michelle Harvie, MD, Principal Investigator — Wythenshawe Hospital
Locations (5):
- United Kingdom (5):
  - Wellcome Trust Clinical Research Facility, Manchester, England
  - Christie Hospital, Manchester, England
  - Nightingale Centre and Genesis Prevention Centre at Wythenshawe Hospital, Manchester, England
  - South Manchester University Hospital, Manchester, England
  - Cancer Care Research Centre at University of Stirling, Stirling, England